CLINICAL TRIAL: NCT02998567
Title: HyPeR: A Phase 1, Dose Escalation Study of Guadecitabine /ASTX727 in Combination With Pembrolizumab (MK3475) in Patients With Refractory Solid Tumours
Brief Title: Combination Study of Guadecitabine/ASTX727 and Pembrolizumab
Acronym: HyPeR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR4420
Record Dates: First submitted 2016-11-02; First posted 2016-12-20 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: immunotherapy; non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — guadecitabine; pembrolizumab; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Escalation (Experimental): Fixed dose of Pembrolizumab with escalating dose of Guadecitabine to establish the phase 2 recommended dose.
  Interventions: Drug: Guadecitabine; Drug: Pembrolizumab
- Expansion (Experimental): Continuation of the Guadecitabine and Pembrolizumab dose established in arm 1: expansion in the recommended patient population.
  Interventions: Drug: Guadecitabine; Drug: Pembrolizumab
- B2: Lung Expansion (Experimental): To further explore the safety and activity of the combination of ASTX727 (replacement of guadecitabine to an oral dose tablet) with pembrolizumab in patients with NSCLC with primary or secondary resistance to PD-1/PD-L1 inhibitors.
  Interventions: Drug: Pembrolizumab; Drug: ASTX727

INTERVENTIONS:
Drug: Guadecitabine — In arm 1 (escalation) and 2 (expansion).
  Arms: Escalation; Expansion
Drug: Pembrolizumab — In arm 1 (escalation) and 2 (expansion).
Drug: ASTX727 — In arm B2 (lung expansion) replacing guadecitabine
  Arms: B2: Lung Expansion

SUMMARY:
HyPeR is a multi-centre Phase 1 Dose Escalation Study of Guadecitabine (SGI-110)/ASTX727 a Second Generation Hypo-Methylating Agent in Combination with Pembrolizumab (MK3475) in Patients with Refractory Solid Tumours. The investigators will be investigating the safety and toxicity of the combination.

DETAILED DESCRIPTION:
This is a multi-centre, dose escalation, Phase I trial. There are two parts to this study. Part A: dose escalation, and Part B: dose expansion.

Part A (Dose Escalation): Patients with advanced solid tumours will be recruited in cohorts of 3 to 6 patients to investigate the combination of 200 mg of pembrolizumab administered as an intravenous injection (first dose given in Cycle 2 Day 8 and then Day 1 of subsequent Cycles) with escalating doses of guadecitabine administered via a subcutaneous injection once a day for 4 days (Days 1-4) of a 21-day cycle.

Once the MTD is reached (or under the advice from the SRC) patients will be enrolled to the dose expansion phase (Part B).

Part B1 (Dose Expansion): 20 patients will be recruited to Part B1 (expansion phase) to further explore the safety and activity of the combination of guadecitabine and pembrolizumab. This cohort will include, but not be limited to, patients with: secondary resistance to PD-1/PD-L1 inhibitors, patients with primary resistance to PD-1/PD-L1 inhibitors in subgroups predicted to benefit such as those with microsatellite-instability high (MSI-H) tumours and/or those with deficient mismatch repair (dMMR) and, possibly other solid tumours based on emerging anti-tumour activity data from Part A and any other relevant preclinical or clinical published data.

Part B2 (NSCLC Dose Expansion): Up to 25 evaluable patients will be recruited to Part B2 (expansion phase) to further explore the safety and activity of the combination of ASTX727 and pembrolizumab. This cohort will include patients with NSCLC with primary or secondary resistance to PD-1/PD-L1 inhibitors. Utilising a Simon's minimax two-stage design, Part B2 will have 80% power with a one-sided significance level of 5% to discount a response rate of 10% in favour of a response rate of 30%. Fifteen patients will be enrolled to stage one, and if two or more patients experience a response (PR or CR by RECIST v1.1), then a further 10 patients will be enrolled to stage two, totaling 25 patients overall.

ELIGIBILITY:
Inclusion Criteria:

1. Part A and B1/2:

   Histologically or cytologically confirmed advanced solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.

   Part B1:

   Histologically or cytologically confirmed advanced solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient AND:
   * Patients with any tumour type that previously responded to a PD-1 or PD-L1 inhibitor and subsequently progressed (defined as secondary resistance to PD-1/PD-L1 inhibitors ie CR or PR by RECIST, or SD by RECIST for 6 months' duration) or/
   * Patients with microsatellite-instability-high (MSI-High) tumours, provided they have been defined by validated assays or patients with deficient mismatch repair (dMMR) defined by immunohistochemistry, who have previously received and have progressed on a PD-1 or PD-L1 inhibitor (primary resistance to PD-1/PD-L1 inhibitors) or/
   * Patients with other solid tumour types who could benefit, based on emerging anti-tumour activity data, from combination therapy with a demethylating agent and PD-1 or PD-L1 inhibitors, in consultation with any other relevant preclinical or clinical data, at the Chief Investigator's discretion.

   Part B2:

   Patients with histologically or cytologically confirmed NSCLC previously treated with PD-1 or PD-L1 inhibitor for advanced or metastatic disease.
2. Life expectancy of at least 12 weeks.
3. Eastern Co-operative Oncology Group (ECOG) performance status of 0-1 with no significant deterioration over the previous 2 weeks (Appendix 1).
4. Evaluable or measurable disease as assessed by RECIST 1.1.
5. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) prior to administration of any investigational medicinal product.

   * Haemoglobin (Hb) ≥ 9.0 g/dL
   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * International normalised ratio (INR) ≤ 1.5x upper limit of normal (ULN)

Or:

Prothrombin time ≤ 1.5x upper limit of normal (ULN)

* Serum bilirubin ≤1.5x ULN

Or:

Direct bilirubin (for patients with total bilirubin >1.5x ULN) ≤ 1.5x ULN

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5x ULN (for patients with liver metastases ≤ 5x ULN is permissible)
* Calculated creatinine clearance (per institutional standard) ≥ 50 mL/min 6.18 years or over. 7. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.

  8. Agree to the use of archival paraffin embedded tissue (if available) for PD-L1 (programmed death-ligand 1) analysis 9. Agree to provide a fresh tumour biopsy at baseline and on Cycle 2 Day 8 of a tumour lesion not previously irradiated (tumours progressing in a prior site of radiation are allowed for PD-L1 characterization, other exceptions may be considered after consultation with the Chief Investigator).

  10. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year. Decitabine, a metabolite of Guadecitabine/ASTX727, can affect fertility and so oocyte cryopreservation should be discussed with female patients.

  12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy. Decitabine, a metabolite of Guadecitabine/ASTX727, can affect fertility and so cryopreservation of sperm should be discussed with male patients.

Exclusion Criteria:

1. Radiotherapy (except brief course for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C and 4 weeks for investigational medicinal products) before treatment, except for hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with CRPC, which are permitted.
2. Patient has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ bladder or cervical cancer that has undergone potentially curative therapy.
3. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
4. Ongoing toxic manifestations of previous treatments. Exceptions to this are:

   * Grade 1 toxicities, which in the opinion of the investigator should not exclude the patient
   * Alopecia of any grade
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the chief Investigator.
6. Has an active autoimmune disease that has required systemic treatment in past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with Sjogren's syndrome will not be excluded from the study. In addition patients that experienced a Grade 2 or higher immune-related AE's on treatment with immunotherapy will be excluded from the study.
7. Has evidence of interstitial lung disease.
8. Has a history of (non-infectious) pneumonitis that required steroid treatment or has active pneumonitis. Pneumonitis includes acute interstitial pneumonitis, pneumonitis and idiopathic pneumonia syndrome.
9. Active infection, requiring systemic therapy.
10. Has received a live vaccine within 30 days of planned start of study therapy. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
11. Major surgery (excluding minor procedures, e.g. placement of vascular access) from which the patient has not yet recovered.
12. At high medical risk because of severe or uncontrolled non-malignant systemic disease including active uncontrolled infection, active bleeding diathesis.
13. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
14. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms (ECGs) within 5 minutes of each other.
    * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete left bundle branch block, third degree heart block.
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
    * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association [NYHA Grade 2 (refer to Appendix 4)]
    * Uncontrolled hypertension - Systolic BP >160mmHg and/or diastolic BP >100mmHg
    * Left ventricular ejection fraction (LVEF) below institutional lower limit of normal.
15. History of hypersensitivity to active or inactive excipients of guadecitabine or pembrolizumab or drugs with a similar chemical structure or class to either agent.
16. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of guadecitabine and pembrolizumab. Participation in an observational trial would be acceptable.
17. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Establish maximum tolerated dose (MTD) | 12 months
  To establish a maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of the combination of guadecitabine and pembrolizumab in patients with advanced solid tumours.
  To determine the maximum dose at which no more than 1 of 6 patients at the same dose level experience a drug related toxicity (DLT), as defined in section 3.1.4 of the protocol.
Measure Adverse Events according to CTCAE v4.0 | 24 months
  To assess the safety and toxicity profile of the combination of guadecitabine and pembrolizumab.
  To determine causality and grading severity of each adverse event by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Pharmacodynamic profile of guadecitabine in combination with pembrolizumab. | 24 months
  Transcriptome analysis in whole bloods using the PAXgene assay.
Pharmacodynamic profile of guadecitabine in combination with pembrolizumab. | 24 months
  Targeted sequencing in plasma circulating free DNA.
Pharmacodynamic profile of guadecitabine in combination with pembrolizumab. | 24 months
  White blood cell analysis by flow cytometry.
Pharmacodynamic profile of guadecitabine in combination with pembrolizumab. | 24 months
  DNA methylation analysis in blood peripheral blood mononuclear cells (PBMC).
Pharmacodynamic studies in guadecitabine in combination with pembrolizumab. | 24 months
  Immunohistochemistry of immune cell in serial biopsies.
Pharmacodynamic studies in guadecitabine in combination with pembrolizumab. | 24 months
  DNA methylation analysis in serial biopsies.
Pharmacodynamic studies in guadecitabine in combination with pembrolizumab. | 24 months
  Transcriptome analysis in serial biopsies.

OTHER OUTCOMES:
Preliminary assessment of the anti-tumour activity | 24 months
  Target lesions will be measured according to RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Marsden Hospital, Sutton, Surrey
  - UCLH, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papadatos-Pastos D, Yuan W, Pal A, Crespo M, Ferreira A, Gurel B, Prout T, Ameratunga M, Chenard-Poirier M, Curcean A, Bertan C, Baker C, Miranda S, Masrour N, Chen W, Pereira R, Figueiredo I, Morilla R, Jenkins B, Zachariou A, Riisnaes R, Parmar M, Turner A, Carreira S, Yap C, Brown R, Tunariu N, Banerji U, Lopez J, de Bono J, Minchom A. Phase 1, dose-escalation study of guadecitabine (SGI-110) in combination with pembrolizumab in patients with solid tumors. J Immunother Cancer. 2022 Jun;10(6):e004495. doi: 10.1136/jitc-2022-004495. PMID 35717027
- See also: Related Info — https://jitc.bmj.com/content/10/6/e004495